CLINICAL TRIAL: NCT00952796
Title: A Comparative Study of Ampicillin/Sulbactam Versus Moxifloxacin in the Treatment of Complicated Intra-abdominal Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Trauma Service Office, kaohsiung medical university hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU-IRB-970389
Record Dates: First submitted 2009-03-01; First posted 2009-08-06 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2009-01

CONDITIONS: Intra-abdominal Infection
Keywords: intra-abdominal infection; moxifloxacin; ampicillin/sulbactam
MeSH Terms: conditions — Intraabdominal Infections | interventions — Moxifloxacin; sultamicillin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): patients with intra-abdominal infection treated with moxifloxacin 400mg once daily
  Interventions: Drug: moxifloxacin
- 2 (Active Comparator): patients with intra-abdominal infection treated with ampicillin/sulbactam 1.5g 4 times daily
  Interventions: Drug: ampicillin/sulbactam

INTERVENTIONS:
Drug: moxifloxacin — moxifloxacin 400mg once daily (IV form, 60minutes)
  Arms: 1
Drug: ampicillin/sulbactam — ampicillin/sulbactam 1.5g 4 times daily (IV form, administered 60minutes)
  Arms: 2

SUMMARY:
On the basis of monotherapy for intra-abdominal infection, the investigators are conducting this study to identify the difference of drug efficacy between ampicillin/sulbactam and moxifloxacin.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed of complicated intra-abdominal infection need surgical treatment

Exclusion Criteria:

* patients diagnosed of intra-abdominal infection receive non-operative management
* patients with known allergic history of fluoroquinolone
* Severe, life threatening disease with a life expectancy of < 48 h or APS and APACHE scores of > 35

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
clinical response at test-of-cure visit | test of cure: 10-14 days after initial treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Department of Emergency Medicine/Surgery, Kaohsiung, Taiwan, Taiwan